CLINICAL TRIAL: NCT02689830
Title: Prostate Embolization for Acute Urinary Retention Study (PARIS 1): An Open-label Prospective Study
Brief Title: Prostate Embolization for Acute Urinary Retention Study
Acronym: PARIS1
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: ClinSearch (Other)
Collaborators: Biocompatibles UK Ltd (Industry); European Georges Pompidou Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SA-112043
Record Dates: First submitted 2016-02-10; First posted 2016-02-24 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Prostatic Hypertrophy, Benign
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bead Block microspheres (Experimental): Prostate embolization
  Interventions: Device: Bead Block

INTERVENTIONS:
Device: Bead Block — Prostate embolization

SUMMARY:
The purpose of this study is to assess the feasibility and safety of Prostate Artery Embolization (PAE) in patients suffering of Acute Urinary Retention (AUR) in the context Benign Prostatic Hypertrophy (BPH).

DETAILED DESCRIPTION:
This is an open-label prospective, multicenter (centralized procedure), single arm, sequentially enrolling study. Twenty subjects will be enrolled in the study.

Patient will be referred by the attending urologists after failure of the currently recommended approach of Trial WithOut Catheter (TWOC) and alpha-adrenergic receptor (AR) blockers.

It is expected that all AUR cases referred to the local urological clinic will be considered for inclusion in the trial. A trial log book will be completed by the referring local urologist in order to obtain preliminary data on the applicability of the trial to all AUR comers in the institution. This log book will be limited to a very simple questionnaire to ensure high rate of completion by the attending resident/fellow (Patients age, size of prostate, previous Benign Prostate Hypertrophy symptoms, renal function). It will be used in order to assess the external validity of this first phase trial and will be a help to design the potential next step trial.

When a patient will present with AUR in the corresponding urological clinic, the PI and Clinical research coordinator will be informed by a short text message, fax or e-mail in order to prepare the following process.

Patient will be informed by the urologist of the ongoing research project. In summary, this will consist in informing the patient that the first step is TWOC and in case of failure of TWOC several options are offered including PAE in the trial setting. Inclusion of the patient will considered only in case of failure of TWOC.

If the patient is willing to participate, patient will be seen in clinic by the Principal Investigator or co-investigator in order to inform him of the protocol and obtain signed informed consent.

PAE will be scheduled upon the first contact to make sure that PAE is performed in a short delay following failure of TWOC. The goal is to perform PAE in the week following recatheterization. For practical reasons this delay might be extended and will be recorded in the Case Report Form.

ELIGIBILITY:
Inclusion Criteria:

* AUR Patients presenting with a first episode of AUR related to BPH (no matter if previously known or not) AND
* Failure of at least one TWOC AND
* Prostate size > or = 50 ml (ultrasound measurement)

Exclusion Criteria:

* Known hypocontractile bladder
* AUR related to other causes (Acute prostatitis or documented Prostate cancer)
* Severe iodine allergy
* Known prostate cancer
* Known ongoing acute or chronic prostatitis
* On-going acute pyelonephritis or septicemia from urinary origin
* Patient refusing PAE
* Severe renal failure (creatinine Clearance < 20 ml/min (MDRD)
* Contra-indication to AR blockers (postural hypotension micturition syncope)
* Contra-indication to anticoagulants
* Patient catheterized with a suspubian catheter
* Patient <18
* Patients who are prisoners
* Patients who are mentally incapacitated
* Patients participating in an investigational study involving the peripheral vasculature
* Patients unable or unwilling to provide written informed consent
* Patients ineligible for pelvic angiography and embolization including severe atheromatous condition or any anatomical condition

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Procedure success | 6 months after PAE
  percentage of patients free of Foley and/or any prostate surgery

SECONDARY OUTCOMES:
Percentage of procedure related or contributed complications | 1 week after PAE
Percentage of immediate technical success of embolization | 5 minutes after the beginning of the procedure
  Percentage of bilateral embolization
Cumulative number of per-procedure angiographic and clinical complications | 24 hours after PAE
  according to the Society of Interventional Radiology and Dindo classifications
Immediate technical success of embolization | 5 minutes after the beginning of the procedure
  percentage of unilateral versus percentage of bilateral embolization
Comparison of International Prostate Symptom Score | between pre-PAE and 3 months post-PAE
Comparison of International Index of Erectile Function | between pre-PAE and 3 months post-PAE
Comparison of Quality of Life Questionnaire | between pre-PAE and 3 months post-PAE
Comparison of International Prostate Symptom Score | between pre-PAE and 6 months post-PAE
Comparison of International Index of Erectile Function | between pre-PAE and 6 months post-PAE
Comparison of Quality of Life Questionnaire | between pre-PAE and 6 months post-PAE
Number of re-catheterization | 6 months after PAE
Time of re-catheterization | 6 months after PAE
Time until TransUrethral Resection of the Prostate or open surgery | 6 months
Cumulative number of days with bladder catheter | between PAE and 6 months post-PAE
Number of patients free of bladder catheter | between PAE and 6 months post-PAE
Number of cumulated hospitalization days | between initial AUR and 6 months post-PAE
Number of cumulated hospitalization days | between PAE and 6 months post-PAE
Total number of consultations | between PAE and 6 months post-PAE
  consultations with interventional radiologist and/or urologist
Prostate volume | 6 months
  Measured with MRI or ultrasound
Comparison of the number of Benign Prostate Hypertrophy medication | before and 3 months after PAE
Comparison of the number of Benign Prostate Hypertrophy medication | before and 6 months after PAE

CONTACTS AND LOCATIONS:
Overall Officials: Marc SAPOVAL, Principal Investigator — HEGP, Paris
Locations (3):
- France (3):
  - Hôpital Saint-Louis, Paris
  - Hôpital Cochin, Paris
  - Hôpital Européen Georges Pompidou, Paris

IPD SHARING:
Plan to Share IPD: Yes
Global results will be available for patients.